CLINICAL TRIAL: NCT07141342
Title: The Fast In-Bed Tracking (FIT) System Lifestyle Intervention
Brief Title: Fast In-Bed Tracking (FIT) System Lifestyle Intervention is a Clinical Trial of a Bed Scale Device. Overweight Wheelchair Users Will Participate in a Weight Loss Program, Half Will Receive Bed Scales, and Participants Who Receive the Bed Scales Are Expected to Have Increased Weight Loss.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Pearlman (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); NuRelm, Inc. (Industry); Craig Hospital (Other)
Responsible Party: Sponsor-Investigator, Jonathan Pearlman, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY24090093; 1R44HD114504-01A1 (NIH)
Record Dates: First submitted 2025-08-13; First posted 2025-08-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Disability Physical; Wheelchair; Obesity; Overweight
Keywords: Wheelchair; Wheelchair Users; Weigh loss; Weight loss device; Weight loss program; device research; bed scale; Wheelchair Scale
MeSH Terms: conditions — Obesity; Overweight | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GLB-AIM (Active Comparator): All participants in the control group will receive the Group Lifestyle Balance Adapted for Individuals with Impaired Mobility (GLB-AIM) intervention. The investigators anticipate a total of 46 participants will be randomized to the control group.
  THE GLB-AIM is a 12-month intervention with a total of 23 sessions: 13 weekly core sessions to start the program, followed by 3 bi-weekly support sessions, and reducing to 1 monthly support session for the final 7 months.
  Control participants will be asked to download the My Net Diary app onto their personal phone and to log daily food intake and exercise using the app for the first 13 weeks of the GLB-AIM program.
  All subjects in the study will be enrolled in the GLB-AIM intervention; the only difference between the experimental and control group is that the control group will not receive the Fast In Bed Tracking System (FIT) scale during the study and therefore will not have the ability to self-monitor their weight.
  Interventions: Behavioral: Group Lifestyle Balance Adapted for Individuals with Impaired Mobility (GLB-AIM) intervention
- GLB-AIM + FIT Weight Scales (Experimental): All participants in the experimental group will receive the Group Lifestyle Balance Adapted for Individuals with Impaired Mobility (GLB-AIM) intervention and will be asked to download the My Net Diary app. The investigators anticipate a total of 46 participants will be randomized to the experimental group.
  Participants who are randomized to the FIT Weight Scale Group will have the FIT scale set up in-home during the baseline visit by research team members. Intervention participants will be oriented to their scale if randomized into the FIT scale group.
  Participants will be asked to enter their weight daily into the My Net Diary app.
  Interventions: Device: The Fast In-Bed Tracking System (FIT) Weight Scale; Behavioral: Group Lifestyle Balance Adapted for Individuals with Impaired Mobility (GLB-AIM) intervention

INTERVENTIONS:
Device: The Fast In-Bed Tracking System (FIT) Weight Scale — It is hypothesized that wheelchair users who are randomized into the FIT Weight Scales group will lose a significantly greater percent of body weight over time (6 months, 12 months) than wheelchair users randomized to the control group.
  Arms: GLB-AIM + FIT Weight Scales
Behavioral: Group Lifestyle Balance Adapted for Individuals with Impaired Mobility (GLB-AIM) intervention — The GLB-AIM is a direct adaptation of the Diabetes Prevention Program (DPP) - Group Lifestyle Balance (DPP-GLB) which has successfully yielded an average 6 percent weight loss at 12 months and reduced diabetes risk over 2.8 years by 58 percent, which was 39 percent lower than participants randomized to the metformin group. The GLB-AIM which has been proven feasible and effective in a pilot study and a randomized control trial (RCT) with 67 mobility impaired individuals randomized to the intervention group or a waitlist control group. There were significant between group differences in weight loss at 6 months (-1.7 kg loss vs 0.05 kg gain, p <0.05) and combined results from both groups after receiving the intervention revealed an average weight loss at 12 months of 3.3 percent of their starting weight. Notably, the average loss was lower than the 5 to 7 percent achieved by diverse participants in the DPP-GLB trials.

SUMMARY:
This project will complete the final design and development steps to commercialize the Fast In-Bed Tracking (FIT) Platform, which is an e-Health and wellness Internet of Things (IoT) monitoring system that can be integrated into a user's bed and provide person-centered, real-world outcomes to support health and wellness. The technical feasibility of FIT was proven over the past several years and has demonstrated the platform can support the treatment of several chronic conditions across different populations, including obesity, congestive heart failure, and pressure injuries. The project goals will be to (1) complete design refinements for FIT and (2) demonstrate the platform's efficacy to support weight loss goals of wheelchair users. Wheelchair users are twice as likely as the general population to be overweight or obese and excess weight not only exacerbates mobility and participation limitations but increases risk for secondary health problems. Evidence reveals that frequent weight monitoring is a key driver for weight management, which puts wheelchair users at a significant disadvantage, because they have no convenient way to measure their body weight. As a recent example, lack of participant's ability to self-weigh was a noted limitation to a weight loss program for wheelchair users, known as the Group Lifestyle Balance weight loss program Adapted for Individuals with Impaired Mobility (GLB-AIM). FIT solves this challenge by passively monitoring a user's weight when they get on and off their bed. The investigators lab and community-based feasibility trials demonstrated that FIT successfully tracks weight for individuals and couples sharing a bed and that users find FIT highly usable. This proposed project will allow the investigators to complete the design refinements participants recommended during our community-based feasibility trial and subsequently examine the efficacy of FIT in supporting the weight-loss goals of community-dwelling wheelchair users through a randomized controlled trial using the GLB-AIM.

DETAILED DESCRIPTION:
Wheelchair users and people with mobility impairments face increased risks of many chronic diseases including hypertension, diabetes, cardiovascular disease, and obesity. Physical inactivity of wheelchair users is related to cardiovascular disease, high blood pressure, diabetes, osteoarthritis, osteoporosis, pressure ulcers, urinary tract infections, and repetitive strain injuries in upper extremities. These health problems cause a downward spiral and are major causes of mortality and morbidity in people with disabilities. This evidence indicates that a physically active lifestyle and healthy weight are critical for people with disabilities, especially wheelchair users, to avoid obesity-related health risks and enjoy a better quality of life.

The World Health Organization (WHO) indicates that worldwide obesity has nearly tripled since 1975. United States data from 2017 to 2020 reveal that 41.9 percent of American adults are obese and estimates indicate that obesity accounts for 173 billion dollars in annual healthcare costs. The distribution of body mass index (BMI) in the country shows 68.8 percent of adults older than 20 years are either overweight or obese.

Wheelchair users have significantly increased risk of obesity and obesity-related health consequences compared to the general population. For instance, Weil et al. found people with lower extremity disabilities to be two and a half times more likely to be obese than the general population. Unfortunately, very little research has been focused on addressing obesity issues for people with disabilities despite the substantial health consequences and costs.

Froehlich-Grobe (co-I on this project) and Lollar state that that "people with disabilities should be an emerging population of concern within public health efforts related to obesity. The three core public health functions of assessment, policy development, and assurance are used as a framework to address this serious public health threat for this group." As part of the policy development section, the authors further state that "research should examine environmental and contextual factors related to physical activity, nutritional intake, and weight maintenance among people with disabilities."

Lifestyle intervention programs exist which address these risks and specific barriers faced by wheelchair users. For individuals with mobility impairments, a host of complex issues make maintaining a healthy weight difficult. Physical barriers to exercise and physical activities, attitudinal barriers towards disability and health, environmental barriers for participation, and challenges with weight monitoring are some of the issues cited by the research community. Further, researchers have noted that individuals with impaired mobility face disability-related challenges that may reduce engagement in programs and interventions. Barriers include transportation and access to travel, caregiver availability to support program engagement, and health-related issues that may prohibit an individual from leaving the home or healthcare setting. These challenges motivated co-I Froehlich-Grobe and colleagues to develop the Group Lifestyle Balance Adapted for Individuals with Impaired Mobility, known as the GLB-AIM. The GLB-AIM is a direct adaptation of the Diabetes Prevention Program (DPP) - Group Lifestyle Balance (DPP-GLB) which has successfully yielded an average 6 percent weight loss at 12 months and reduced diabetes risk over 2.8 years by 58 percent, which was 39 percent lower than participants randomized to the metformin group. The GLB-AIM which has been proven feasible and effective in a pilot study and a randomized control trial (RCT) with 67 mobility impaired individuals randomized to the intervention group or a waitlist control group. There were significant between group differences in weight loss at 6 months (-1.7 kg loss vs 0.05 kg gain, p <0.05) and combined results from both groups after receiving the intervention revealed an average weight loss at 12 months of 3.3 percent of their starting weight. Notably, the average loss was lower than the 5 to 7 percent achieved by diverse participants in the DPP-GLB trials.

The effectiveness of these programs for wheelchair users is hampered by the lack of a self-management strategy which most of the population takes for granted: a weight monitoring tool.

A crucial difference between the DPP-GLB and GLB-AIM trials is the weekly self-monitoring of weight as a form of accountability. In the DPP-GLB programs participants are weighed by the intervention coaches at the weekly meetings, which was not possible to do in the GLB-AIM as one disability-specific adaptation made to reduce transportation barriers to participation was that sessions were delivered telephonically most weeks, with participants only coming in once a month for an in-person session during which their weight would be obtained. But as most participants do not have accessible scales at home, they were unable to assess their weight weekly. Self-weighing frequency is associated with significantly greater weight loss, weight maintenance, and less body mass.

Evidence suggests that over a two-year period individuals who self-weigh daily will lose up to 18 lbs. more than those who do not self-weigh as frequently, and individuals who self-weigh more frequently are 60 to 80 percent more likely to maintain their weight. Unfortunately people with mobility impairments who are unable to stand or have balance issues do not have technology that is feasible for them to use to self-weigh frequently, which has been a noted limitation of weight loss interventions for this population.

Most wheelchair users do not have accessible scales at home and few primary health care providers have accessible scales to weight their patients who use wheelchairs. In fact, a recent survey of over 700 US physicians revealed that less than a quarter (22.6 percent) reported using an accessible scale to measure weight, while 72 percent relied on asking the patient to self-report their weight. Our colleague and co-investigator on this project, Dr. Froehlich-Grobe, reported that the average amount of time that had passed since wheelchair users in a previous trial had been weighed was 19.6+41.4 months, which suggests that most wheelchair users do not have an accurate estimate of their weight.

Although internet-enabled scales are available for in-home that range in price from 50 to 200 dollars, no equivalent technology exists for wheelchair users who cannot stand. Hospital and clinic-based scales such as roll-on, lift-based, and integrated bed scales are available for weight measurement but have little applicability in the home. Roll-on scales, for instance, are expensive, too large for most homes, and require the person to be weighed in their wheelchair and then transferred out of the wheelchair so that the wheelchair can be weighed separately, which makes self-weighing difficult without assistance. Lift-based scales are also large, expensive, and require assistance since the wheelchair user must be transferred onto the lift's platform for weighing. Hospital-based bed scales are convenient for the in-patient population but are not applicable for in-home use for several reasons: they cannot be integrated into a user's current bed; they do not accommodate weight measurement for multiple people (e.g. husband/wife); they are expensive; they do not provide the affordance of monitoring with mobile devices; and there is evidence that they are not accurate. Consequently, if wheelchair users want to monitor their weight, they often schedule a visit to the clinic or simply estimate their weight which is known to be inaccurate. The need for an easy-to-use home-based scale motivated us to develop the Fast In-Bed Tracking System (FIT).

The FIT will provide wheelchair users with an accurate, affordable, practical weight monitoring system. The investigators propose work to support refinements and translation of the FIT, which is a low-cost, easy-to-use scale that can be integrated into any bed which will automatically log weight for wheelchair users who use a bed without changes to their daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Age18 +
* Live within approximately 75 miles of Pittsburgh
* Uses a wheelchair as primary means of locomotion
* Currently transfers in and out of bed every night (or most nights)
* Has been diagnosed as obese or overweight
* Are interested in losing weight
* BMI in the range of approximately 25 to 40; BMI range will be determined from published evidence for the primary diagnosis of the participant. For example, spinal cord injury /quadriplegic BMI range of approximately 22 to 40; for amputees it will be based on location and level of amputation, or if no diagnosis specific evidence exists, a BMI of approximately 25 to 40 will be used as a general guideline.
* Own a smart phone, and have reliable internet and wifi connection
* Are comfortable using exercise equipment like resistance bands or hand pedal exercisers
* Are able and willing to engage in exercise of moderate intensity
* Weight in bed including sleep partner is an estimated combined weight of 600 pounds or less
* Does not have a regular way to weigh themselves, such as a roll-on scale in the home or gym, or have regular access to a device to weigh themselves regularly and are willing to avoid weighing themselves during the trial.
* Indication that the participant has autonomy in decision-making as determined by the "Everyday Autonomy Self-Determination Scale."
* Indication that their current bedroom setup is compatible with the FIT bed scales as determined by the "Bed Determination Survey."

Due to the medical complexity of this population, inclusion of this study based on BMI, in-bed transfer frequency, or geographic location will be at the discretion of the expert members of our study team and will be considered on a case-by-case basis.

Exclusion Criteria:

* Extended vacations or absences planned in the next year (more that 2 - 4 weeks) or plans to move approximately 75 miles or greater from the Pittsburgh region
* BMI outside of the desired range as based on condition and as determined by the study team.
* Currently taking weight loss medication, medications that affect appetite, or have had weight loss surgery in the last 2 years.
* History disordered eating in the last 2 years, such as Anorexia Nervosa, Bulimia Nervosa or Binge Eating Disorder
* Currently pregnant or intend to become pregnant in the next 12 months
* Regularly have 4 or more alcoholic drinks a day
* Have any cognitive conditions that limit decision making or self-governing.
* Indication that the participant does not have autonomy in decision-making as determined by the "Everyday Autonomy Self-Determination Scale."
* Indication that their current bedroom setup is not compatible with the FIT bed scales as determined by the "Bed Determination Survey."

Due to the medical complexity of this population, exclusion from this study based on BMI, geographic location, and what is considered a "medication that affects appetite" will be at the discretion of the expert members of our study team and will be considered on a case-by-case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Weight Loss after 6 and 12 months comparing the intervention group (FIT bed scale with daily weight feedback) versus control group (weighed at baseline, 6 and 12 months) | Baseline, Month 6, Month 12
  The difference in weight loss from baseline to 6 and 12 months (intervention versus control groups).

SECONDARY OUTCOMES:
Participant's Adherence to the Diet and Exercise Intervention (Average Days Per Week of Food Tracking) | Baseline to Month 12
  MyNetDiary food intake entries will be collected from the participant's MyNetDiary account. Adherence to daily food tracking will be reported as average days per week of food tracking.
Participant's Average Daily Caloric Intake when Tracking Food | Baseline to Month 12
  MyNetDiary food intake entries will be collected from the participant's MyNetDiary account on a weekly basis. Daily caloric intake when tracking food will be calculated by dividing the total amount of calories consumed in the week by the number of days in the week participant's tracked food.
Changes in Participant's Body Composition | Baseline, Month 6, Month 12
  Waist Circumference is measured using a tailor's measuring tape, measuring the waist circumference of the participant (just above the navel) in centimeters.
Changes in Participant's Dietary Intake | Baseline, 6 and 12 months
  Changes in dietary intake will be recorded via a 3-day recall using the Automated Self-Administered Dietary Assessment Tool (ASA-24). Targeted categories will include: Total Calories, Fat, Protein, Fruit, and Vegetables.
Average weekly minutes of physical activity (strength, aerobic) | Baseline to Month 12
  Daily exercise (minutes and type of exercise) will be entered into the MyNetDiary App, specifically strength and aerobic activity. Average minutes of exercise per week will be reported.
Usability and acceptability of the Fast In-Bed Tracking (FIT) bed scale | Months 1, 6 and 12
  A questionnaire on the usability and acceptability of the FIT bed scale will be completed by participants. The form integrates free-text questions to participants on the usability of the software, hardware and appearance of the FIT bed scale with a standardized System Usability Scale (SUS). The SUS is a 10 question form with a 5 answer rating scale of Strongly Disagree - Strongly Agree, weighted 1 - 5 points respectively. Odd numbered questions are calculated by subtracting 1 from the participant response. Even numbered questions are calculated by subtracting the participant response from 5. The converted responses are added up and multiplied by 2.5, which converts the range of possible values from 0 to 100. Higher scores indicate a more positive perception of the device, with an average score being about 68.
Changes in Participant's Sleep Duration and Quality | Baseline, 6 and 12 months
  Sleep duration and quality changes will be reported via the Brief Pittsburgh Sleep Quality (B-PSQI) questionnaire. Changes in sleep quality and duration are linked to a healthy diet and exercise, and these metrics are being collected to understand participant's changes in sleep quality in relation to the diet and exercise intervention as a projection of overall health outcomes. There are 6 questions that participants will answer about their average sleep in the previous month: time to bed, time getting up, time taken to fall asleep, duration of their sleep, frequency of waking up the night, and an overall rating of their sleep quality. There are 5 scorable items in a range of 0 - 3 , as bed time and rise time are combined to create a single score (Greater than 7 hours equals zero, less than 5 hours equals 3) to create a global score with a range of 0 - 15. Higher scores indicate worse sleep quality.
Changes in Participant's Self-Efficacy in Health Practices | Baseline, 6 and 12 months
  The Self-Rated Abilities for Health Practices Scale (SRAHP) is a questionnaire used to assess an individual's perceived ability to engage in health-promoting behaviors. It consists of 28 items across four subscales: Nutrition, Psychological Well-being, Exercise, and Responsible Health Practices. Each item is rated on a 5-point Likert scale of 0 to 4, with 0 representing "not at all" and 4 representing "completely", with higher scores indicating greater self-perceived ability. Scoring: Individual subscale scores are calculated by summing the ratings for each item within that subscale. The total score is the sum of all subscale scores. The total score ranges from 0 to 112, with higher scores reflecting greater self-efficacy for health practices.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Pearlman, PhD, Principal Investigator — University of Pittsburgh; Katherine Froehlich-Grobe, PhD, Study Director — Craig Hospital
Locations (1):
- University of Pittsburgh, Bakery Square, Department of Rehabilitation Science and Technology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as a condition of IRB approval and individual experiences of the clinical trial will not be of clinical relevance to the field. Aggregate data will be released as to the efficacy of the device to be studied in the clinical trial.

REFERENCES:
- See also: This is the participant-facing ASA-24 where they will complete their dietary recalls. — https://asa24.nih.gov/
- See also: This is the website attached to the app that participants will download to their phones to complete dietary recall for intervention purposes. Researchers can invite participants into specified groups. — https://www.mynetdiary.com/